CLINICAL TRIAL: NCT00107874
Title: Oral Misoprostol as a Second-line Alternative to Intravenous Oxytocin in Preventing Postoperative Blood Loss After Non-scheduled Cesarean Section: a Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Oral Misoprostol Versus Intravenous Oxytocin in Preventing Blood Loss After Non-scheduled Cesarean Section
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: M73/99
Record Dates: First submitted 2005-04-11; First posted 2005-04-12 (Estimated); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Postpartum Hemorrhage
Keywords: Maternal; morbidity; mortality; pregnancy; postpartum hemorrhage; Cesarean Section
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: misoprostol

SUMMARY:
Postpartum hemorrhage (PPH) ranks among the leading causes of maternal morbidity and mortality, both in developed and developing countries.

With this trial, we sought to determine the effectiveness of oral misoprostol as an uterotonic drug in comparison with intravenous oxytocin, in patients with a low risk of PPH undergoing non-scheduled Cesarean section.

We therefore compared the intra- and postoperative blood loss, as well as drug related side effects in patients, treated by the same surgical and anesthesiological team in one institution.

DETAILED DESCRIPTION:
Postpartum hemorrhage (PPH) is still among the leading causes of maternal morbidity and mortality. The incidence of PPH is reduced by active management of the third stage of labor which includes the use of uterotonics for pharmacological prophylaxis. However, there is an on-going debate about the optimal drug selection since uterotonics such as oxytocin and methylergometrine are liable for specific side effects and complications when administered within a dose range needed to be effective for PPH. In the search for an alternative to these conventional standard uterotonics, misoprostol (prostaglandin E1) has turned out to be an effective therapeutic option and has been implemented in actual treatment regimens. The objective of this study was to compare the effectiveness of oral applicated misoprostol versus intravenous oxytocin in reducing blood loss in low risk obstetric patients undergoing non-scheduled cesarean section (CS) under spinal anesthesia.

Comparison:

In this prospective, double blind study, parturients undergoing CS were randomized to receive either a) oral misoprostol and an infusion of normal saline supplemented with placebo, or b) an oral placebo and an infusion of normal saline, supplemented with oxytocin subsequently to intravenous oxytocin after cord clamping in both groups.

The primary outcomes were the amount of intra- and postoperative blood loss and the occurrence of drug-related side effects.

ELIGIBILITY:
Inclusion Criteria:

* Non-scheduled primary or secondary Cesarean section (CS) after the 37th week of gestation

Exclusion Criteria:

* Emergency CS
* Fetal distress
* Fetal malformations
* Preeclampsia and HELLP (Hemolysis-Elevated Liver enzymes-Low Platelet count syndrome)
* Hypersensitivity to prostaglandins
* Coagulopathy
* Severe systemic disorders
* An American Society of Anesthesiologists (ASA) physical status >/= 3
* Severe asthma
* Prior myomectomy
* Maternal fever (> 38.5 °C)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 1999-01; Primary Completion 2002-02 (Actual); Study Completion 2002-02 (Actual)

PRIMARY OUTCOMES:
Reduction of postpartum hemorrhage

SECONDARY OUTCOMES:
Blood loss
medicamentous side effects
efficacy of medicaments

CONTACTS AND LOCATIONS:
Overall Officials: Irène Hösli, Prof. Dr. MD, Study Chair — University Hospital, Basel, Switzerland
Locations (1):
- Women's University Hospital, Basel, Basel, Switzerland